CLINICAL TRIAL: NCT03413241
Title: Pain in Autism Spectrum Disorder (ASD): A Psychophysical and Neurophysiological Exploration of Pain Sensitivity and Its Relation to Clinical Characteristics
Brief Title: Pain in Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: ASD 0496-17-RMB
Record Dates: First submitted 2018-01-21; First posted 2018-01-29 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: High-functioning Autism
Keywords: autism spectrum disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The proposed project will be first performed on individuals with HF-ASD with their expected heterogeneity and healthy control (HC) subjects in order to explore the pain processing and modulation mechanisms underlying the pain sensitivity profile of adults with HF-ASD. Secondly, we will focus on individuals with ASD and HC, without ASR (ASD-nonASR, HC-nonASR) and with SHR (ASD-SHR, HC-SHR). This 2X2 factorial design will enable us to determine whether the feature of SHR in individuals with HF-ASD contributes to pain sensitivity. This research project will comprise of two sessions. Session I will include the following tests ADOS-2 for ASD diagnosing (only for individuals with ASD), intelligence quotation testing (IQ Wechsler Abbreviated Scale of Intelligence® - Second Edition (WASI®-II)107, serving for inclusion criteria. Session II will include familiarization with the researchers and lab, thermal detection threshold testing for small fiber abnormality identification since detection thresholds in some reports found to be abnormal pain threshold testing, and completion of questionnaires (see section 3.6 for details), psychophysical testing and EEG recordings in the following order: i) rEEG recordings; ii) psychophysical pain assessments; simultaneously with iii) neurophysiological pain assessments with pain EPs recorded. Our research protocol will be approved by the Helsinki Committee of the Rambam Health Care Center and The Chaim Sheba Medical Center.

DETAILED DESCRIPTION:
A dysregulation of the balance between excitatory and inhibitory neural activity (i.e. an E/I imbalance) underlies ASD pathology. Neural hyper-responsiveness and impaired top-down modulation represent the E/I imbalance, underpinning the ASD clinical characteristics. One of the most frequent ASD characteristics is atypical sensory responsiveness, including exaggerated behavioral responses to sensory stimuli (i.e. sensory hyper-responsiveness). In healthy subjects, sensory hyper-responsiveness was found to be associated with pain hyper-sensitivity.This study project aims to study whether : (1) the individuals with ASD exhibit pain hyper-sensitivity, namely a pro-nociceptive profile, supported by the E/I imbalance. (2) the pain sensitivity will be positively associated with ASD clinical characteristics, and (3) sensory hyper-responsiveness will be found to be a contributing factor to pain hyper-sensitivity in ASD individuals.

We will perform a multi-method, comprehensive psychophysical and neurophysiological evaluation of pain sensitivity along with self-reports of clinical characteristics, daily function, and quality of life. The participants will be high functioning ASD (HF-ASD) individuals (IQ >80). Pain processing by means of pain hyperalgesia and pain inhibition capability, along with EEG activity at rest and in response to noxious stimuli (pain-evoked potentials), will be compared between ASD subjects and healthy controls. The best pain-related psychophysical and/or neurophysiological measures differentiating between groups will be tested for correlations with the ASD clinical characteristics. In order to test the contributing role of sensory hyper-responsiveness to pain sensitivity in ASD, the aforementioned psychophysical and neurophysiological evaluation will be performed in 4 homogenous groups: ASD with and without sensory hyper-responsiveness, and controls with and without sensory hyper-responsiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Proficiency in using the Hebrew language;
2. Verbal performance and full scale estimate of 80 and above on the WASI
3. No use of pain medication for the past 24 hours.
4. Inclusion criteria for the ASD group: A diagnosis of HF-ASD based on the ADOS-2

Exclusion Criteria:

1) Diagnosis of chronic pain.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: 80 adults (18-45 years) diagnosed with HF-ASD, and up to 92 healthy subjects, controlled for age, sex and IQ,
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2018-05-06 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Pain processing and modulation mechanisms underlying the pain sensitivity profile of adults with HF-ASD | 4 years
  To explore the pain processing and modulation mechanisms underlying the pain sensitivity profile of adults with HF-ASD

CONTACTS AND LOCATIONS:
Locations (1):
- The lab of clinical neurophysiology, the faculty of medicine, Technion and Rambam Medical Center, Haifa, Israel